CLINICAL TRIAL: NCT02406014
Title: Efficacy and Safety of Ingenol Mebutate Gel 0.015% Compared to Diclofenac Sodium Gel 3% in Subjects With Actinic Keratoses on the Face or Scalp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LP0041-1120
Record Dates: First submitted 2015-03-27; First posted 2015-04-01 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2017-05

CONDITIONS: Actinic Keratosis (AK)
MeSH Terms: conditions — Keratosis, Actinic | interventions — 3-ingenyl angelate; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group A (Active Comparator): Ingenol mebutate gel 0.015%, once daily for 3 consecutive days for the first treatment course. At 8 weeks after treatment initiation, subjects who present with existing AKs or newly emergent AKs in the treatment area will receive one more treatment course of ingenol mebutate gel 0.015%, daily for 3 consecutive days.
  Interventions: Drug: Ingenol Mebutate Gel, 0.015%
- Treatment Group B (Active Comparator): Diclofenac sodium gel 3%, (0.5 grams), twice daily for 90 days.
  Interventions: Drug: Diclofenac sodium gel 3%

INTERVENTIONS:
Drug: Ingenol Mebutate Gel, 0.015% — Ingenol mebutate gel 0.015 % (Picato®) applied on the selected treatment area. Retreatment if the treatment field is not completely cleared of AKs.
  Other Names: Picato®
  Arms: Treatment Group A
Drug: Diclofenac sodium gel 3% — Diclofenac sodium gel 3% Solaraze® applied on the selected treatment area, twice daily for 90 days.
  Other Names: Solaraze®
  Arms: Treatment Group B

SUMMARY:
This is a phase 4, multi-centre, randomized, two group, open label, active controlled, parallel group, 17 week trial.

DETAILED DESCRIPTION:
All subjects who qualify for this trial are to have 4 to 8 clinically typical, visible and discrete AK lesions within a contiguous 25 cm2 treatment area on the face or scalp.

Eligible subjects will be randomised in a 1:1 ratio to the following treatment groups:

* Treatment Group A: Ingenol mebutate gel 0.015%, once daily for 3 consecutive days for the first treatment course. At 8 weeks after treatment initiation, subjects who present with existing AKs or newly emergent AKs in the treatment area will receive one more treatment course of ingenol mebutate gel 0.015%, daily for 3 consecutive days.
* Treatment Group B: Diclofenac sodium gel 3%, (0.5 grams), twice daily for 90 days.

ELIGIBILITY:
Inclusion Criteria:

1. Following verbal and written information about the trial, subject must provide informed consent documented by signing the Informed Consent Form (ICF) prior to any trial related procedures
2. Subjects with 4 to 8 clinically typical, visible and discrete AKs within a contiguous 25 cm² treatment area on the face or scalp

Exclusion Criteria:

1. Location of the selected treatment area:

* on the periorbital skin
* on the perioral skin/around the nostrils
* within 5 cm of an incompletely healed wound
* within 10 cm of a suspected BCC or SCC or other neoplasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Complete clearance of all AKs | 11 Months
  Complete clearance of all AKs in the treatment field at Week 8 for ingenol mebutate gel 0.015% and Week 17 for diclofenac sodium gel 3%

SECONDARY OUTCOMES:
Complete clearance of all AKs at Week 17 | 11 Months
  As secondary response criteria, complete clearance at Week 17 for diclofenac sodium gel 3% will be compared with complete clearance in the ingenol mebutate 0.015% group.

CONTACTS AND LOCATIONS:
Overall Officials: Eggert Stockfleth, Prof.Dr.med., Principal Investigator — St. Josef-Hospital im Katholischen Klinikum Bochum
Locations (1):
- Gemain, Weber & Craninic, Schweinfurt, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stockfleth E, Harwood CA, Serra-Guillen C, Larsson T, Osterdal ML, Skov T. Phase IV head-to-head randomized controlled trial comparing ingenol mebutate 0.015% gel with diclofenac sodium 3% gel for the treatment of actinic keratosis on the face or scalp. Br J Dermatol. 2018 Feb;178(2):433-442. doi: 10.1111/bjd.16048. Epub 2018 Jan 15. PMID 29030864